CLINICAL TRIAL: NCT01157442
Title: Harnessing Mobile Phone Usage for HIV and Horizontal Health Systems Improvement: PMTCT
Brief Title: Study of Cell Phone SMS Messages for Prevention of Maternal to Child Transmission of HIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: University of Nairobi (Other); Canadian International Development Agency (Other Government)
Responsible Party: Dr. Joshua Kimani, University of Manitoba and UNiversity of Nairobi
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H2009:315
Record Dates: First submitted 2010-07-02; First posted 2010-07-07 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2010-07

CONDITIONS: HIV Infections
Keywords: prevention of maternal to child transmission of HIV; mhealth; access to antenatal care; pregnancy
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cell phone sms messages (Experimental): The experimental arm will receive the cell phone SMS text messaging intervention.
  Interventions: Behavioral: cell phone sms text messaging
- Control (No Intervention): The control group will receive the standard of care but no SMS text messages.

INTERVENTIONS:
Behavioral: cell phone sms text messaging — At enrollment a study nurse will send the intervention group a weekly SMS message reminding them to attend antenatal care. Starting at 36 weeks gestational age, an automated bulk SMS management system, will send the intervention group 3 SMS text messages (using non descript slogans) each week by proxy reminding them to take their nevirapine in labor. From time of delivery to 6 weeks postpartum the women will aslo receive 3 SMS messages per week reminding them to attend their 6 week checkup and 6 week infant visit.Upon receiving these messages women in the intervention group can text back if they have any concerns or questions. These women would then receive phone calls from the study nurse triaged according to the women's needs.
  Arms: cell phone sms messages

SUMMARY:
Optimal development of sustainable health systems must use locally relevant infrastructure. Mobile phone technology, driven primarily by local market forces rather than foreign assistance, is spreading rapidly through African communities to improve people's personal and business communications. Here, the investigators propose using a structured mobile phone communications system for prevention of mother to child transmission of HIV (PMTCT). The system is designed to improve antenatal linkage to care, provide reminders to take PMTCT medications, and improve post-natal support and follow-up, even when mothers deliver at home. In addition to benefits in PMTCT related outcomes, this model allows evaluation of the intervention in a public health setting with the ultimate goal of advancing regional health systems development. The overall goal of of the study is to assess if mobile phones and SMS text messages can be used to help improve prevention of maternal to child transmission (PMTCT) of HIV services by strengthening health systems.

Specific objectives are:

1. To determine if mobile phone SMS text messages can demonstrate an improvement in compliance with a known intervention ( use of nevirapine) for PMTCT, demonstrated by:

1a) improved antenatal care attendance (greater than 4 visits)

1b) increased usage of nevirapine in labour (from 60% to at least 70%)

1c) earlier identification and treatment of HIV positive infants

1d) increased postpartum care for HIV positive mothers

1e) acceptability of cell phone SMS text messages transmission of information among HIV positive women

2. To demonstrate that mobile phone technology can be used as an effective tool to strengthen PMTCT health information systems at the facility level by: 2a) determining factors that constrain or promote the use of cell phone technology to strengthen PMTCT health information systems from the perspective of patients, health care providers and policy makers 2b) determining how cell phones can be used as a tool to generate equity statistics for PMTCT programs and formulate equity orientated PMTCT policies 2c) determine if early involvement of policy makers in the study improves knowledge translation

ELIGIBILITY:
Inclusion Criteria:

Women will be eligible to participate if they:

* are pregnant with a singleton pregnancy,
* attend care at Pumwani Maternity Hospital,
* are HIV positive,
* have never had a preterm birth (before 37 weeks),
* are planning to reside in Nairobi for at least 6 months post delivery,
* live within 15 km of PMH,
* have basic literacy skills in Kiswahili or English,
* are willing to be contacted for follow up and have their own cell phone or regular access to their partners' cell phone (partners must be aware of their HIV status).

Exclusion Criteria:

* Women who are pregnant and attend care at Pumwani Maternity Hospital who are not HIV positive,
* Women who have had a preterm birth,
* Women who are not planning to reside in Nairobi for at least 6 months post delivery,
* Women who do not live within 15 km of PMH,
* Women who do not have basic literacy skills in English or Kiswahili
* Women who are not willing to be contacted for follow up,
* Women who do not have their own cell phone or regular access to their partner's cell phone and
* Women whose partner's are not aware of their HIV status.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 856 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
increased nevirapine uptake in labour in pregnant HIV positive women from 60% to 70% | At time of delivery and/or postpartum visit

SECONDARY OUTCOMES:
HIV positive rates in infants born to mothers in the study | assessed at birth, 6 weeks and 3 months of age
number of antenatal care visits | assessed at time of 6 week postpartum visit
earlier identification and treatment of HIV positive infants | at 6 week infant visit
acceptability fo smsm messages for PMTCT related care | at 6 week postpartum visit

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Kimani, MD, Principal Investigator — University of Manitoba and University of Nairobi; Peter Cherutich, MD, Principal Investigator — Ministry of Health, NASCOP Kenya; Mary Gichuihi, Masters, Study Director — University of Nairobi
Locations (1):
- Pumwani Maternity Hospital, Nairobi, Kenya